CLINICAL TRIAL: NCT04522141
Title: Testing Self-Control as a Behavior Change Mechanism to Increase Physical Activity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Margie Lachman, Minnie and Harold Fierman Professor of Psychology, Brandeis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20100R; 5P30AG048785 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Sedentary Lifestyle; Self-control
Keywords: Physical exercise; Behavior change
MeSH Terms: conditions — Sedentary Behavior; Self-Control; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-control treatment group (Experimental): The self-control treatment group will wear a Fitbit step counter across 8 weeks. In addition, they will use the MindHike smartphone application across 8 weeks. Each day, the app sends the a reminder to wear the Fitbit as well as a short interventional input targeting self-control.
  Interventions: Behavioral: Self-control intervention
- Control group (Active Comparator): The control group will wear a Fitbit step counter across 8 weeks. In addition, they will use the MindHike smartphone application across 8 weeks. Each day, the app sends the a reminder to wear the Fitbit.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Self-control intervention — Participants will wear a Fitbit for 8 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. Across the 8 weeks, participants receive daily reminders to wear their Fitbit. After the baseline week, participants will also receive interventional components that target self-control via the smartphone application MindHike. This intervention should help them achieve their activity goals. The self-control intervention teaches strategies how to potentiate desirable impulses and how to avoid undesirable impulses in daily life.
  Arms: Self-control treatment group
Behavioral: Control condition — Participants will wear a Fitbit for 8 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. Participants in this condition receive daily reminders to wear their Fitbit through the MindHike smartphone application. Participants in the control group will be matched with the self-control intervention group for how much contact they have with the app and the researchers.
  Arms: Control group

SUMMARY:
The goal of this study is to test self-control as a behavior change mechanism for physical activity and to investigate whether a smartphone-based self-control intervention can increase physical activity among sedentary middle-aged adults.

DETAILED DESCRIPTION:
It is widely known that being physically active is beneficial for one's health and well-being, yet only a small percentage of adults engage in the recommended amounts of physical activity. Research has shown that health-damaging behaviors such as a sedentary lifestyle can be attributed in part to a lack of self-control. There is some evidence that self-control strategies can be improved with targeted interventions. The overall aim of the proposed study is to test self-control as a behavior change mechanism for physical activity and to investigate whether a smartphone-based self-control intervention can increase physical activity among sedentary middle-aged and older adults. To test the effect of this self-control intervention, participants will be randomized into two conditions: The self-control treatment group and the control group. Both groups will track their daily physical activity using a Fitbit step counter over eight weeks. Additionally, the self-control intervention group will receive a 7-week smartphone-based self-control intervention to learn strategies how to potentiate desirable impulses or weaken undesirable ones. It is expected that the self-control treatment group will show greater increases in physical activity and that changes will last longer compared to the control group. Self-control is expected to mediate the relationship between condition and physical activity. It is predicted that the self-control treatment group will show greater changes in self-control compared to the control group and that people who increase more in self-control also increase more in their physical activity. Two versions of the MindHike smartphone application will be used to communicate with all participants. The self-control treatment group will receive a version delivering a self-control intervention. The control group will receive a minimal version without the interventional components. Both groups are matched in terms of contact frequency.

ELIGIBILITY:
Inclusion Criteria:

* between 35-65 years of age
* fluent in English
* fit enough to walk for at least 20 min at a time
* owns a smartphone

Exclusion Criteria:

* experienced a fall or heart problem/condition in the last 6 months
* is currently participating in an exercise program to increase physical activity
* is already physically active (physically active = exercise regularly 3 times per week, or more for at least 30min)
* was advised by a doctor to not walk due to health conditions

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margie Lachman, PhD, Principal Investigator — Brandeis University
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stieger M, Allemand M, Lachman ME. Effects of a digital self-control intervention to increase physical activity in middle-aged adults. J Health Psychol. 2023 Sep;28(10):984-996. doi: 10.1177/13591053231166756. Epub 2023 Apr 12. PMID 37042306
- [Derived] Stieger M, Allemand M, Lachman ME. Targeting self-control as a behavior change mechanism to increase physical activity: Study protocol of a randomized controlled trial. Contemp Clin Trials. 2021 Jan;100:106236. doi: 10.1016/j.cct.2020.106236. Epub 2020 Dec 1. PMID 33276145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-control Treatment Group | Control Group
Started | 42 | 39
Completed | 41 | 39
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant did not complete the baseline (pretest) but provided activity data.
  Not all participants answered all questions/questionnaires because they were allowed to skip questions hence the discrepancy between measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-control Treatment Group | Control Group | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.90 (7.16) | 49.24 (11.28) | 46.96 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 29 | 62
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 38 | 38 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 27 | 30 | 57
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: Objective Physical Activity
Description: Average daily steps baseline week, average daily steps between pretest and posttest, and average daily steps between posttest and followup. A higher score means more steps.
Time Frame: Average daily steps baseline week (week 1); average daily steps between pretest and posttest (week 2-8); average daily steps between posttest and followup (week 9-12)
Population: Please note that some participants did not answer all questions/questionnaires because they were allowed to skip questions hence the discrepancy between measures. Some participants did not provide their step data.
Measure: Mean (Standard Deviation); unit: Average Daily Steps
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 37 | 38
Average Daily Steps
  Average daily steps baseline week (week 1) | 6184.45 (3084.61) | 6671.81 (4213.50)
  Average daily steps between pretest and posttest (weeks 2-8) | 6647.71 (2787.96) | 6932.25 (6071.56)
  Average daily steps between posttest and follow-up (weeks 9-12): number analyzed (Participants) | 35 | 35
  Average daily steps between posttest and follow-up (weeks 9-12) | 6426.23 (3167.05) | 6722.13 (4638.01)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.038, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.941, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

2. Primary Outcome: Self-Reported Physical Activity
Description: International Physical Activity Questionnaire - short version. A continuous score will be calculated expressed as MET (Metabolic Equivalents) minutes per week: Total MET-min/week = (Walk METs*min*days) + (Mod METs*min*days) + Vig METs*min*days). A higher score means higher level of physical activity.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: Please note that some participants did not answer all questions/questionnaires because they were allowed to skip questions hence the discrepancy between measures.
Measure: Mean (Standard Deviation); unit: MET minutes/week
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 38 | 33
MET minutes/week
  T1 | 1598.95 (2461.04) | 2460.11 (4157.84)
  T2 | 3268.70 (3754.73) | 3122.72 (3811.26)
  T3 | 3891.36 (6362.59) | 2778.18 (3586.78)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.003, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.027, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

3. Primary Outcome: Self-Control
Description: The Brief Self-Control Scale was used to measure self-control. Items are assessed from 1 (not at all) to 5 (very much). A mean across all items will be calculated. A higher score means a higher score in self-control.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale
  T1 | 3.32 (0.60) | 3.42 (0.75)
  T2 | 3.54 (0.63) | 3.62 (0.76)
  T3 | 3.63 (0.65) | 3.63 (0.75)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p < .001, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.411, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

4. Primary Outcome: Weekly Self-Control
Description: The Brief Self-Control Scale was used to measure weekly self-control. Items are assessed from 1 (not at all) to 5 (very much). A mean across all items will be calculated. A higher score means a higher score in self-control. Participants were asked to answer the items with respect to the last week.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 41 | 36
units on a scale
  Week 1 | 5.81 (1.31) | 6.28 (1.48)
  Week 2 | 6.07 (1.50) | 6.14 (1.66)
  Week 3 | 6.11 (1.51) | 6.52 (1.52)
  Week 4 | 6.26 (1.32) | 6.37 (1.61)
  Week 5 | 6.13 (1.40) | 6.53 (1.56)
  Week 6 | 6.49 (1.30) | 6.52 (1.55)
  Week 7 | 6.53 (1.49) | 6.46 (1.44)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect weekly self-control; Test type: Other; p < .001, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction weekly self-control; Test type: Superiority; p = 0.176, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

5. Secondary Outcome: Big Five Personality Traits
Description: The Big Five Inventory 2 was used to assess the Big Five personality traits. Items are assessed from 1 (disagree strongly) to 5 (agree strongly). A mean across all items per personality trait will be calculated. A higher score means a higher score on a personality trait.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale
  T1 Extraversion | 3.41 (.72) | 3.34 (.86)
  T2 Extraversion | 3.49 (.65) | 3.43 (.87)
  T3 Extraversion | 3.44 (.68) | 3.35 (.93)
  T1 Agreeableness | 3.95 (.62) | 3.89 (.66)
  T2 Agreeableness | 3.90 (.59) | 3.85 (.63)
  T3 Agreeableness | 3.70 (.63) | 3.78 (.63)
  T1 Conscientiousness | 3.87 (.72) | 3.90 (.80)
  T2 Consientiousness | 3.92 (.66) | 3.89 (.81)
  T3 Conscientiousness | 3.88 (.67) | 3.78 (.71)
  T1 Neuroticism | 2.82 (.91) | 2.90 (1.00)
  T2 Neuroticism | 2.80 (.88) | 2.82 (.89)
  T3 Neuroticism | 2.76 (.89) | 2.83 (.94)
  T1 Open-Mindedness | 4.07 (.54) | 4.04 (.82)
  T2 Open-Mindedness | 3.93 (.69) | 4.05 (.76)
  T3 Open-Mindedness | 3.92 (.63) | 3.99 (.82)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p > .05, Mixed Models Analysis — Analyses are controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p > .05, Mixed Models Analysis — Analyses are controlled for age, sex, education, race, self-reported functional health, and self-reported health status

6. Secondary Outcome: Exercise Self-efficacy
Description: Nine items were used to assess how sure participants are that they will exercise under certain circumstances (e.g., when you are feeling under pressure or when you are away from home). Items were assessed from 1 (very sure) to 4 (not at all sure). A mean across all items will be calculated. A higher score means lower exercise self-efficacy.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 37
units on a scale
  T1 | 2.43 (.89) | 2.48 (.95)
  T2 | 2.33 (.78) | 2.15 (.80)
  T3 | 2.26 (.81) | 2.14 (.74)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.031, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.260, Mixed Models Analysis; Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

7. Secondary Outcome: Satisfaction With Life
Description: The Satisfaction with life scale was used to assess satisfaction with life. Items were assessed from 1 (disagree strongly) to 7 (agree strongly). A mean across all items will be calculated. A higher score means a higher satisfaction with life.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale
  T1 | 4.55 (1.40) | 4.00 (1.49)
  T2 | 4.64 (1.57) | 4.24 (1.61)
  T3 | 4.75 (1.41) | 4.08 (1.58)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.016, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.363, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

8. Secondary Outcome: Sense of Control
Description: 12 items were used to assess sense of control. The scale consisted of two subscales: personal mastery (e.g., I can do just about anything I really set my mind to) and perceived constraints (e.g., What happens in my life is often beyond my control). All items were rated on a scale ranging from strongly agree (1) to strongly disagree (7). All items were coded so that a higher score reflected greater personal mastery and greater perceived constraints, respectively.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale
  T1 Personal Mastery | 5.64 (1.20) | 5.75 (1.27)
  T2 Personal Mastery | 5.59 (1.08) | 5.66 (1.03)
  T3 Personal Mastery | 5.75 (.98) | 5.41 (1.32)
  T1 Perceived Constraints | 3.33 (1.35) | 3.23 (1.34)
  T2 Perceived Constraints | 3.35 (1.44) | 3.32 (1.43)
  T3 Perceived Constraints | 3.25 (1.52) | 3.48 (1.44)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p > .05, Mixed Models Analysis — Analyses are controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p > .05, Mixed Models Analysis — Analyses are controlled for age, sex, education, race, self-reported functional health, and self-reported health status

9. Secondary Outcome: Stop & Go Switch Task
Description: To measure attention switching and inhibitory control, we used the newly developed online app version of the Stop & Go Switch Task (SGST). The SGST requires alternating between the "normal" condition (i.e., respond "Go" to the stimulus "Green" and "Stop" to the stimulus "Red") and the "reverse" condition (i.e., respond "Stop" to the stimulus "Green" and "Go" to the stimulus "Red"). For the SGST, the total number of correct responses across the mixed trials were calculated. Total range: 0 - 32. A higher score means a better outcome.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 41 | 36
score on a scale
  T1 | 27.32 (3.07) | 24.72 (7.48)
  T2 | 24.08 (6.19) | 25.14 (6.30)
  T3 | 26.46 (4.20) | 25.44 (4.53)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.389, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.516, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

10. Secondary Outcome: Backward Digit Span Test
Description: To measure working memory capacity, we used the backward digit span test from the WAIS-III. The task includes increasingly longer series of digits, ranging from two to eight digits. Participants attempt to repeat them in the reverse order from which they were shown. The score is the longest string that is repeated exactly in reverse order. Digits are presented at a rate of one per second, beginning with a set size of two digits and progressing to eight digits. The accuracy score is the largest set size that was correctly reproduced. Possible range: 0 - 8. A higher score means a better outcome.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
score on a scale
  T1 | 5.17 (2.84) | 4.63 (2.81)
  T2 | 4.30 (3.13) | 4.17 (2.66)
  T3 | 4.11 (3.50) | 3.11 (3.06)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.005, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.555, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

11. Secondary Outcome: Immediate Word List Recall Task
Description: Immediate episodic memory for verbal materials are tested using free recall of a word list drawn from the Rey Auditory-Verbal Learning Test. Participants are instructed to read carefully a list of 15 words which are presented at a rate of one second per word, and then to recall as many words as possible. In scoring the accuracy measure, one point is given for each correct response. Possible range: 0 - 15. A higher score means a better outcome.
Time Frame: Baseline (Pretest) T1, Week 8 (Posttest) T2, Week 12 (Follow-up) T3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-control Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
score on a scale
  T1 | 7.57 (3.17) | 5.84 (2.58)
  T2 | 6.84 (2.44) | 6.69 (3.37)
  T3 | 7.42 (2.70) | 7.41 (2.80)
Statistical Analysis 1: Comparison: Self-control Treatment Group vs Control Group; Main effect; Test type: Other; p = 0.206, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status
Statistical Analysis 2: Comparison: Self-control Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = 0.026, Mixed Models Analysis — Controlled for age, sex, education, race, self-reported functional health, and self-reported health status

ADVERSE EVENTS:
Time Frame: 3 months
Description: [Not specified]
Arm/Group | Self-control Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT04522141/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT04522141/ICF_001.pdf